CLINICAL TRIAL: NCT02391818
Title: The Effect of Taxane Chemotherapy on Balance in Breast Cancer Patients
Acronym: IPMR Balance
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Collaborators: Illinois CancerCare, P.C. (Other); University of Illinois College of Medicine at Peoria (Other); St. Francis Hospitals & Health Centers (Other)
Responsible Party: Principal Investigator, Catherine Horst, Principle Investigator, Physical Therapist, OSF Healthcare System
Other Study IDs: 599231-1
Record Dates: First submitted 2015-02-20; First posted 2015-03-18 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Distorted; Balance; Quality of Life; Neuropathy; Cancer
Keywords: balance; quality of life; chemotherapy; neuropathy; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast Cancer Patients receiving ACT: Adraimycin/Cytoxan/Taxol
- Breast Cancer patients receiving RT only: radiation therapy

SUMMARY:
The purpose of this study is to quantify the balance impairments during and after taxane chemotherapy. Disability due to balance impairments caused by chemotherapy induced peripheral neuropathy (CIPN) can cause falls, injury, and a decline in independence. This results in poor treatment outcomes such as greater morbidity and mortality, inability to complete treatment protocols, self-limitation of activity, and diminished quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to describe the balance deficits prior to the initiation of taxane therapy and through the duration of treatment and compare balance to a cohort of women without taxane therapy. To our knowledge, a study like this has not been done yet it is a necessary next step in order to evaluate whether balance deficits resolve independent of treatment or if the balance deficits require targeted therapy. Other studies evaluating balance in taxane patients, have used cross-sectional study designs that are limited to observation at one point in time. Further, other evaluations have been limited in the measurement of balance using only self-report questionnaires, with no performance measurements of functional balance. Previous studies of other conditions have shown poor concordance between self-report questionnaires and performance measures. Therefore, our proposed longitudinal study improves the current knowledge about balance deficits during taxane therapy by quantifying the impact of taxane chemotherapy on balance during and after treatment using standardized and validated self-report and performance functional balance assessment tools. The results of this study will improve the treatment of balance deficits in women with taxane therapy by identifying the type, onset, duration, and severity of the deficits within each balance system. From these findings, targeted interventions, if required, could be developed. In addition, establishing feasibility and utility for quantifying balance impairments is necessary for the development of larger studies assessing the effects of rehabilitation interventions on functional disability due to CIPN. Such a study would be worthy of influencing changes in clinical practice to minimize disability from balance dysfunction before, during, and after chemotherapy, and thus maximizing function and quality of life during and after cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women with breast cancer (stage 0-III)
2. Scheduled to receive any of the following individual treatment protocols:

   1. ACT
   2. Radiation only

Exclusion Criteria:

1. Required assistive device for ambulation in the 6 months prior to starting treatment
2. Previous taxane or platinum chemotherapy (paclitaxel/Taxol®, docetaxel/Taxotere®, cabazitaxel/Jevtana®, cisplatin, carboplatin, and oxaliplatin)
3. Inability to stand or walk without assistance
4. BMI >40 (see chart below)
5. Pre-existing vestibular, visual, somatosensory, orthopedic, and neurologic disease before entering the study including but not limited to being legally blind (ICD9 368.3, 369.0-369.2 lower extremity amputation (ICD9 895.0-897.7), and Diabetes (ICD9 249.0-250.93, 257.2)
6. Evidence of central nervous system metastasis
7. Cognitive difficulties or medical conditions that, in the opinion of the study investigators, will affect testing protocols
8. Enrollment in other trial aimed at treating CIPN.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from cancer treatment clinic and radiation oncology clinics
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline Modified Clinical Test of Sensory Integration of Balance at 9 months. | An average of 5 months for the controls, and 9 months for the cases.
  assessment of static balance under conditions eyes open on firm surface, eyes closed on firm surface, eyes open on foam surface, and eyes closed on foam surface

SECONDARY OUTCOMES:
Change from baseline Five Times Sit to STand | An average of 5 months for the controls, and 9 months for the cases.
  Time in seconds it takes to stand up and sit down from a standard height chair
Change from baseline Visual Contrast Sensitivity | An average of 5 months for the controls, and 9 months for the cases.
  Using the Mars Letter Chart, a contrast sensitivity score is calculated
Change from baseline Touch Detection Threshold | An average of 5 months for the controls, and 9 months for the cases.
  The lightest Von Frey Filament able to be detected using the up/down method is recorded on 3 places of each foot
Change from baseline Patient Neurotoxicity Questionnaire | An average of 5 months for the controls, and 9 months for the cases.
  Likert scale describing the level of intensity of lower extremity neuropathy symptoms and their interference with functional activities
Change from baseline Patient Neuropathy Function Questionnaire | An average of 5 months for the controls, and 9 months for the cases.
  number of falls are recorded, as well as Likert scales for various functional activities
Change from baseline Edmonton Symptom Assessment Scale | An average of 5 months for the controls, and 9 months for the cases.
  Quality of life scale validated for the breast cancer population

CONTACTS AND LOCATIONS:
Overall Officials: Carl Asche, PhD, Study Director — University of Illinois College of Medicine at Peoria; Jinma Ren, PhD, Study Director — University of Illinois College of Medicine at Peoria; Catherine Horst, DPT, Principal Investigator — IPMR; Nguyet Le-Lindqwister, MD, Study Director — Illinois CancerCare; Anthony Zalduendo, MD, Study Director — OSF Radiation Oncology
Locations (4):
- United States (4):
  - Illinois CancerCare, Pekin, Illinois
  - OSF Radiation Oncology, Pekin, Illinois
  - Illinois CancerCare, Peoria, Illinois
  - OSF Radiation Oncology, Peoria, Illinois

REFERENCES:
- [Background] Wampler MA, Topp KS, Miaskowski C, Byl NN, Rugo HS, Hamel K. Quantitative and clinical description of postural instability in women with breast cancer treated with taxane chemotherapy. Arch Phys Med Rehabil. 2007 Aug;88(8):1002-8. doi: 10.1016/j.apmr.2007.05.007. PMID 17678662
- [Background] Winters-Stone KM, Torgrimson B, Horak F, Eisner A, Nail L, Leo MC, Chui S, Luoh SW. Identifying factors associated with falls in postmenopausal breast cancer survivors: a multi-disciplinary approach. Arch Phys Med Rehabil. 2011 Apr;92(4):646-52. doi: 10.1016/j.apmr.2010.10.039. Epub 2011 Mar 2. PMID 21367394
- [Background] Tofthagen C, Overcash J, Kip K. Falls in persons with chemotherapy-induced peripheral neuropathy. Support Care Cancer. 2012 Mar;20(3):583-9. doi: 10.1007/s00520-011-1127-7. Epub 2011 Mar 5. PMID 21380613
- [Background] Whitney SL, Wrisley DM, Marchetti GF, Gee MA, Redfern MS, Furman JM. Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther. 2005 Oct;85(10):1034-45. PMID 16180952
- [Background] Lord SR, Menz HB. Visual contributions to postural stability in older adults. Gerontology. 2000 Nov-Dec;46(6):306-10. doi: 10.1159/000022182. PMID 11044784
- [Background] Shimozuma K, Ohashi Y, Takeuchi A, Aranishi T, Morita S, Kuroi K, Ohsumi S, Makino H, Mukai H, Katsumata N, Sunada Y, Watanabe T, Hausheer FH. Feasibility and validity of the Patient Neurotoxicity Questionnaire during taxane chemotherapy in a phase III randomized trial in patients with breast cancer: N-SAS BC 02. Support Care Cancer. 2009 Dec;17(12):1483-91. doi: 10.1007/s00520-009-0613-7. Epub 2009 Mar 28. PMID 19330359
- [Background] Hausheer FH, Schilsky RL, Bain S, Berghorn EJ, Lieberman F. Diagnosis, management, and evaluation of chemotherapy-induced peripheral neuropathy. Semin Oncol. 2006 Feb;33(1):15-49. doi: 10.1053/j.seminoncol.2005.12.010. PMID 16473643
- [Background] Dougherty BE, Flom RE, Bullimore MA. An evaluation of the Mars Letter Contrast Sensitivity Test. Optom Vis Sci. 2005 Nov;82(11):970-5. doi: 10.1097/01.opx.0000187844.27025.ea. PMID 16317373
- [Background] Mancini M, Horak FB. The relevance of clinical balance assessment tools to differentiate balance deficits. Eur J Phys Rehabil Med. 2010 Jun;46(2):239-48. PMID 20485226